CLINICAL TRIAL: NCT02571855
Title: Double-blind, Placebo-controlled, Randomized Study to Investigate the Tolerability, Safety, Pharmacokinetics, and Pharmacodynamics of ACT-541468: Part A: Multiple-ascending Doses in Healthy Young Adults After Morning Administration Part B: Single-ascending Doses in Healthy Elderly Subjects After Morning Administration Part C: Repeated Doses in Both Healthy Young Adults and Elderly Subjects After Evening Administration
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of ACT-541468 in Healthy Young Adults and Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AC-078-102
Record Dates: First submitted 2015-10-02; First posted 2015-10-08 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects
Keywords: insomnia; Pharmacokinetics; Safety; Pharmacodynamics; Healthy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — daridorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A: ACT-541468 multiple ascending doses (Experimental): Six young adults will receive ACT-541468 in the morning from Day 1 to Day 5 at each dose level in a sequential manner (total number of subjects = 18). Planned dose levels are 10, 25 and 75 mg per day
  Interventions: Drug: ACT-541468 (hydrochloride salt)
- Part A: Placebo (Placebo Comparator): For each ACT-541468 dose level tested in Part A, 2 young adults will receive matching placebo in the same conditions (total number of subjects = 6)
  Interventions: Drug: Placebo
- Part B: ACT-541468 single ascending doses (Experimental): Six elderly will receive ACT-541468 in the morning of Day 1 at each dose level in a sequential manner (total number of subjects = 18). Planned dose levels are 5, 15 and 25 mg
  Interventions: Drug: ACT-541468 (hydrochloride salt)
- Part B: Placebo (Placebo Comparator): For each ACT-541468 dose level tested in Part B, 2 elderly will receive matching placebo in the same conditions (total number of subjects = 6)
  Interventions: Drug: Placebo
- Part C: repeated dose of ACT-541468 (Experimental): Sixteen young adults and eight elderly will receive ACT-541468 (planned dose: 25 mg) in the evening for 7 days (8 days for 6 of the 16 young adults).
  Interventions: Drug: ACT-541468 (free base)
- Part C: Placebo (Placebo Comparator): Four young adults and 2 elderly will receive matching placebo in the same conditions as subjects receiving the active compound in Part C
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACT-541468 (hydrochloride salt) — Hard-gelatin capsules (strength: 5 mg and 25 mg)
  Arms: Part A: ACT-541468 multiple ascending doses; Part B: ACT-541468 single ascending doses
Drug: ACT-541468 (free base) — Soft capsules (strength: 25 mg)
  Arms: Part C: repeated dose of ACT-541468
Drug: Placebo — Placebo capsules matching the ACT-541468 formulations
  Arms: Part A: Placebo; Part B: Placebo; Part C: Placebo

SUMMARY:
The purpose of this study is to evaluate the tolerability, safety, pharmacokinetics (PK, or amount of drug over time in the body) and pharmacodynamics (PD, or effects on the body) of ACT-541468 following multiple ascending doses in healthy adults and following single ascending doses in healthy elderly subjects when administered in the morning. The safety, PK and PD of ACT-541468 will also be assessed after repeated evening administration of a selected dose in both healthy adults and elderly.

DETAILED DESCRIPTION:
In the first-in-man study, single doses of ACT-541468 administered in healthy young adults were well tolerated up to the dose level of 200 mg (inclusive) and yielded results compatible with possible sleep facilitating effects of ACT-541468. So the present study aimed to further investigate the effects of ACT-541468 after multiple ascending doses in healthy young subjects as well as after single ascending doses in elderly subjects (morning administrations). The effects of repeated administrations of a selected dose administered in the evening in both healthy adults and elderly, will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Adults aged from 18 to 45 years (inclusive) for Part A; elderly aged from 65 to 80 years (inclusive) for Part B; both adults from 18 to 45 years and elderly from 65 to 80 years (inclusive) for Part C.
* Regular sleep pattern of at least 6 hours nocturnal sleep.
* Young females must have negative pregnancy tests at screening and at pre-dose on Day 1 and use a reliable method of contraception
* Body mass index (BMI) between 18.0 and 30.0 kg/m2 (inclusive) at screening.
* Systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate (PR) between 100-145 mmHg, 50-90 mmHg and 45-90 bpm (all inclusive) for young adults, respectively; SBP, DBP and PR between 100-160 mmHg, 50-95 mmHg and 45-100 bpm (all inclusive) for elderly, respectively.
* Healthy on the basis of physical examination,electrocardiogram and laboratory tests.

Exclusion Criteria:

Principal exclusion criteria common to young adults and elderly:

* Pregnant or lactating women.
* Any contraindication to the study drugs.
* History or presence of any disease or condition or treatment, which may put the subject at risk of participation in the study or may interfere with the absorption, distribution, metabolism or excretion of the study drugs.
* History of narcolepsy or cataplexy or modified Swiss narcolepsy scale total score < 0 at screening.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol.

Exclusion criteria for young adults only:

* Treatment with any prescribed medications or over-the-counter medications within 2 weeks prior to study drug administration.

Exclusion criteria for elderly only:

* Previous chronic treatment with any medication that is not given in stable doses and/or stable regimen within 2 months prior to screening.
* Previous treatment with CNS-active drugs or within 2 months prior to screening.
* Treatment with inhibitors of CYP3A4 (e.g., azole derivatives, ritonavir, clarithromycin) from 2 weeks prior to screening visit and up to EOS.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | up to 72 hours post dosing
  Treatment emergent adverse events and treatment emergent serious adverse events will be evaluated throughout the study
Changes from baseline in ECG variables and vital signs (heart rate and blood pressure) | up to 72 hours post dosing
  12-lead electrocardiogram variables including RR, PR, QRS, QT and QTc intervals at scheduled time points during Parts A, B and C
Changes from baseline in clinical laboratory parameters | up to 72 hours post dosing
  Laboratory tests including hematology, blood chemistry and urinalysis at scheduled time points during PArts A, B and C

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of ACT-541468 after daytime and bedtime intake | Part A: Day 1 and Day 5; Part B: Day 1; Part C: evening of Day 8 (pre-dose) and Day 9 (nighttime samples)
  Cmax will be determined after single (Parts A and B) and multiple morning doses (Part A) as well as after repeated evening doses to identify the nighttime PK profile (Part C)
Time to reach Cmax (tmax) of ACT-541468 after daytime and bedtime intake | Part A: Day 1 and Day 5; Part B: Day 1; Part C: evening of Day 8 (pre-dose) and Day 9 (nighttime samples)
  tmax will be determined after single (Parts A and B) and multiple morning doses (Part A) as well as after repeated evening doses to identify the nighttime PK profile (Part C)
Terminal half-life [t(1/2)] after daytime and bedtime intake | Part A: Days 1 and 5, from pre-dose up to 72 h post-dose; Part B: Day 1, at pre-dose up to 72 h post-dose; Part C: from the morning of Day 8 up to 60 h post-dose and from the evening of Day 8 (pre-dose) until 36 h post-dose (with nighttime samples)
  t(1/2) will be determined after single (Parts A and B) and multiple morning doses (Part A) as well as after repeated evening doses (Part C)
Areas under the plasma concentration-time curves [AUC(0-8), AUC(0-24)] of ACT-541468 after daytime and bedtime intake | Part A: Days 1 and 5, from pre-dose up to 72 h post-dose; Part B: Day 1, at pre-dose up to 72 h post-dose; Part C: from the morning of Day 8 up to 60 h post-dose and from the evening of Day 8 (pre-dose) until 36 h post-dose (with nighttime samples)
  AUC from time 0 to 8 hours after study drug administration [AUC(0--8)] and from time 0 to 24 hours after study drug administration [AUC(0--24)] will be determined after single (parts A and B) and multiple morning doses (Part A) as well as after multiple evening doses (Part C)
Areas under the plasma concentration-time curves [AUC(0-t), AUC(0-inf)] of ACT-541468 after daytime and bedtime intake | Part A: Day 5, from pre-dose up to 72 h post-dose; Part B: Day 1, at pre-dose up to 72 h post-dose; Part C: from the morning of Day 8 up to 60 h post-dose and from the evening of Day 8 (pre-dose) until 36 h post-dose (with nighttime samples)
  AUC from time 0 to infinity [AUC(0--inf], AUC from time 0 to time of the last measured concentration above the limit of quantification [AUC(0--t)] will be determined after single (Part B) and multiple morning doses (Part A) as well as after multiple evening doses (Part C)
Sedation as measured by saccadic peak velocity | Part A: Day 1 and Day 5; Part B: Day 1; Part C: Day 2 and Day 14
  saccadic eye movements (SEM) will be recorded by electrooculography and the average values of saccadic peak velocity of the SEM will be used as parameter of sedation
Visual motor coordination | Part A: Day 1 and Day 5; Part B: Day 1; Part C: Day 2 and Day 14
  Visual motor coordination will be assessed with the adaptive tracking test and the average tracking performance will be used as parameter of coordination
Change from baseline in body sway | Part A: Day 1 and Day 5; Part B: Day 1; Part C: Day 2 and Day 14
  Body sway will be assessed using a body sway meter
Change from baseline in subjective cognitive effects | Part A: every day from Day 1 to Day 6; Part B: Day 1; Part C: Day 1 to Day 8
  Subjects will rate sleepiness, alertness and mood using questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Mühlan, MSc, Study Director — Actelion
Locations (1):
- Investigator Site, Leiden, Netherlands

REFERENCES:
- [Derived] Muehlan C, Boehler M, Brooks S, Zuiker R, van Gerven J, Dingemanse J. Clinical pharmacology of the dual orexin receptor antagonist ACT-541468 in elderly subjects: Exploration of pharmacokinetics, pharmacodynamics and tolerability following single-dose morning and repeated-dose evening administration. J Psychopharmacol. 2020 Mar;34(3):326-335. doi: 10.1177/0269881119882854. Epub 2019 Oct 23. PMID 31642731